CLINICAL TRIAL: NCT00938574
Title: A Prospective, Open-label, Single Center, Dose Finding Phase I-study With Atu027 (an siRNA Formulation) in Subjects With Advanced Solid Cancer
Brief Title: Study With Atu027 in Patients With Advanced Solid Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Silence Therapeutics GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Atu027-I-01; EudraCT-No: 2008-005588-32
Record Dates: First submitted 2009-07-13; First posted 2009-07-14 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2012-09

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — Atu027

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Drug Atu027 (Experimental)
  Interventions: Drug: Atu027

INTERVENTIONS:
Drug: Atu027

SUMMARY:
This is a phase I, prospective, open-label, single center, dose finding study with Atu027 (an siRNA formulation) given as single treatment followed by repeated treatment (repeated treatment phase: 8 treatments within 4 weeks) as therapy in subjects with advanced solid cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically and/or cytologically proven advanced, recurrent or metastatic solid malignancy for which standard curative or palliative measures do not exist, are no longer effective, or are unlikely to be effective.
2. Age >/= 18 years.
3. ECOG performance score of 0-2.
4. Life expectancy of at least 3 months.
5. Subjects must have recovered from the acute reversible effects of previous anti-cancer therapies. At least 30 days since major surgery and at least 5 half-lives (t1/2) must have elapsed since treatment with any investigational agent.
6. Adequate marrow, hepatic, renal, and heart function at the time of screening.
7. Weight >/= 50kg.
8. Subjects must have at least one measurable lesion according to RECIST.
9. Women of childbearing potential must have a negative urine pregnancy test at baseline.
10. Women of childbearing potential and men must be willing to use highly effective contraceptive methods during the course of the study and three months after.
11. Subjects must be willing and able (in the opinion of the investigator) to understand the subject information and informed consent form and to comply with the study protocol and procedures.
12. Subjects must be willing and able to give written informed consent.

Exclusion Criteria:

1. Evidence of central nervous system (CNS) metastases.
2. Peripheral venous access insufficient to permit intravenous infusion or acquisition of laboratory specimen.
3. Major surgery within 30 days prior to first study treatment.
4. Evidence that subject has only insufficiently recovered from the acute reversible effects of previous anti-cancer therapies or surgery.
5. Abnormal hematologic parameters as defined:

   * Neutrophil count < 1.500/mm3 (=1.5x10^9/l)
   * Platelet count < 100.00/mm3 (=100x10^9/l)
   * White blood cells < 3x10^9/l
   * Hemoglobin < 9.0 g/l
6. Abnormal renal or hepatic function as defined:

   * ASAT (SGOT), ALAT (SGPT) >/= 1.5xULN or >/= 2.0xULN in case of liver metastases
   * Total bilirubin >/= 1.5xULN
   * Creatinine clearance < 50ml/min calculated by the Cockroft-Gault formula
7. Weight < 50 kg.
8. Any concurrent disease, medical or social condition that could affect compliance with the protocol or interpretation of results as judged by the investigator. In particular, subjects with the following conditions are not allowed to enter the study:

   * Seizures
   * Poorly controlled Diabetes mellitus
   * Lipid metabolism disorder (cholesterol and triglycerides >/= 1.5xULN), Refsum disease
   * Myocardial infarction within six (6) months prior to enrollment or having insufficient cardiac function defined as NYHA Grade 3 or 4, uncontrolled angina, cardiomyopathy, severe uncontrolled ventricular arrhythmias, left bundle branch block or electrocardiographic evidence of acute ischemic or active conduction system abnormalities (e.g. long QT interval, Torsade de Pointes)
   * Poorly controlled hypertension
   * Severe dyspnea or severe pulmonary dysfunction
   * Autoimmune and inflammatory disease
   * Active infection or known bacteremia
   * Known infection with HIV or chronic infection with hepatitis B or C virus
   * History of acute or chronic pancreatitis
   * Substance abuse
9. Prior gene transfer therapy.
10. Concurrent treatment with investigational or commercial agents or therapies administered with the intention to treat the subject's malignancy.
11. Participation in any other clinical study or use of investigational device(s) during participation in this study.
12. Known hypersensitivity to ingredients of the infusion solution.
13. Pregnant or nursing women or women of childbearing potential who are not willing to use highly effective forms of contraception during participation in this study and at least three months thereafter.
14. Male subjects with partners of child-bearing potential who are not willing to use highly effective contraception during participation in this study and for at least three months thereafter, unless surgically sterile.
15. Subject is a relative of, or staff directly reporting to the investigator or employee of the sponsor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2009-06; Primary Completion 2012-07 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Determination of dose-limiting toxicities (DLT) and maximum tolerated dose (MTD) of single and repeated intravenous infusion with Atu027 in subjects with advanced solid tumors | treatment and follow up

SECONDARY OUTCOMES:
Collection of data concerning pharmacokinetics of Atu027 and its components | treatment and follow up
Collection of data concerning clinical safety and tolerability | treatment and follow up
Clinical response as measured by RECIST criteria | treatment and follow up

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Strumberg,, MD, Prof., Director, Principal Investigator — Dept. of Hematology & Med. Oncology, Univ. of Bochum, Marienhospital Herne
Locations (1):
- Dept. of Hematology & Med. Oncology, Univ. of Bochum, Marienhospital Herne, Herne, Germany

REFERENCES:
- [Derived] Schultheis B, Strumberg D, Santel A, Vank C, Gebhardt F, Keil O, Lange C, Giese K, Kaufmann J, Khan M, Drevs J. First-in-human phase I study of the liposomal RNA interference therapeutic Atu027 in patients with advanced solid tumors. J Clin Oncol. 2014 Dec 20;32(36):4141-8. doi: 10.1200/JCO.2013.55.0376. Epub 2014 Nov 17. PMID 25403217